CLINICAL TRIAL: NCT02127476
Title: A Phase 1 Double-blind, Placebo-controlled, Single- and Multiple-ascending-dose Study of KHK6640 in Alzheimer's Disease
Brief Title: A Study of Single and Multiple Doses of KHK6640 in Subjects With Prodromal or Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6640-001; 2013-002873-23 (EudraCT Number)
Record Dates: First submitted 2014-04-24; First posted 2014-04-30 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KHK6640 (Experimental): KHK6640
  Interventions: Drug: KHK6640
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: KHK6640 — Single ascending dose and multiple ascending doses administration
  Arms: KHK6640
Drug: Matching Placebo — Single ascending dose and multiple ascending doses administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of KHK6640, given as a single dose and as multiple doses in patients with Prodromal Alzheimer's Disease (AD) or Mild to Moderate AD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prodromal AD or mild to moderate AD
* Clinical Dementia Rating (CDR) score of 0.5, 1.0, or 2.0
* Have a cognitive impairment
* Low Aβ and high Tau in Cerebrospinal fluid (CSF)
* Mini Mental State Examination (MMSE) score > 16 at Screening

Exclusion Criteria:

* Previous active treatment with an AD immunotherapy in an investigational study
* Use of another investigational drug within 30 days of screening
* History or presence of clinically significant seizures, brain trauma, transient ischemic attack, and/or cerebrovascular disease
* Presence of a neurological condition that could be contributing to cognitive impairment above and beyond that caused by the subject's AD
* Evidence of infection, tumor, or other clinically significant lesions that could indicate a dementia diagnosis other than AD

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-07; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 7 months
  Safety assessment variables will include all adverse events (AEs) including serious and non-serious AEs, laboratory parameters (hematology, chemistry, and urinalysis), vital signs, 12-lead electrocardiograms, physical and neurological examinations, and brain MRI

CONTACTS AND LOCATIONS:
Locations (9):
- UZ Gent, De Pintelaan 185, Ghent, Belgium
- Clinical Research Services Turku (CRST), Itäinen Pitkäkatu 4B,, Turku, Finland
- Netherlands (2):
  - Department of Neurology and Alzheimer Center, VU University Medical Center, Amsterdam
  - University Medical Centre Groningen (UMCG), Alzheimer Research Centre, Groningen
- Serbia (2):
  - Clinical Centre of Serbia, Neurology Clinic, Dr Subotica Starijeg 6 ,, Belgrade
  - Military Medical Academy, Crnotravska 17,, Belgrade
- Sweden (3):
  - Memory Clinic, Malmo Minneskliniken, Memory Research Unit, Hs 33,, Malmo
  - Sahlgrenska Gothenburg, Minnesmottagningen, Wallinsgatan 6, Mölndal
  - Karolinska Stockholm Karolinska University Hospital, Huddinge, Dept. of Geriatrics/Memory Disorders Unit, Stockholm